CLINICAL TRIAL: NCT01901575
Title: Remifentanil IV PCA for Ablation of Idiopathic Ventricular Tachycardia
Brief Title: Remifentanil Intravenous Patient Controlled Analgesia (IVPCA) for Ablation of Idiopathic Ventricular Tachycardia
Acronym: IVPCA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-00800
Record Dates: First submitted 2013-04-16; First posted 2013-07-17 (Estimated); Results first posted 2014-12-19 (Estimated); Last update posted 2018-01-02 (Actual); Status verified 2017-12

CONDITIONS: Tachycardia, Ventricular
Keywords: idiopathic ventricular tachycardia
MeSH Terms: conditions — Tachycardia, Ventricular | interventions — Remifentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Remifentanil IV PCA (Experimental): patients with PVC's prior to administration of remifentanil
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Remifentanil — Patients with established PVC's , sedated with remifentanil IVPCA per study protocol
  Other Names: Ultiva

SUMMARY:
Determine effects of remifentanil conscious sedation in patients undergoing Electrophysiological (EP) studies for the ablation of idiopathic ventricular tachycardia and/or persistent frequent premature ventricular contractions (PVCs) of non-ischemic origin

DETAILED DESCRIPTION:
The purpose of the study is to determine the effects of remifentanil conscious sedation in patients undergoing Electrophysiological (EP) studies for the ablation of idiopathic ventricular tachycardia and/or persistent frequent PVCs of non-ischemic origin.

Remifentanil is an analgesic- synthetic opiate with an very short half life. It is rapidly broken down by enzymes in the blood and is ideally suited for continuous sedation. The effect is practically eliminated within 5 minutes after the intravenous sedation is stopped.

You are being asked to participate in this study because you are already scheduled to undergo EP studies under the care of your cardiologist for the ablation of idiopathic ventricular tachycardia and/or persistent frequent PVCs of non-ischemic origin.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo EP studies for the ablation of idiopathic ventricular tachycardia and/or persistent frequent PVCs of non-ischemic origin
* Patients between 18 and 65
* ASA 1-3

Exclusion Criteria:

* ASA 4 and 5
* Age 18 and 65

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Misha Kogan, MD, Principal Investigator — NYU School of Medicine
Locations (1):
- NYU Langone Medical Center, New York, New York, United States

REFERENCES:
- [Background] Garofalo NA, Teixeira-Neto FJ, Schwartz DS, Vailati Mdo C, Steagall PV. Effects of the opioid remifentanil on the arrhythmogenicity of epinephrine in halothane-anesthetized dogs. Can J Vet Res. 2008 Jul;72(4):362-6. PMID 18783026

RESULTS

PARTICIPANT FLOW:
Groups:
- Remifentanil IV PCA: Patients with established PVC's sedated with remifentanil IVPCA per study protocol
Period: Overall Study
Arm/Group | Remifentanil IV PCA
Started | 16 (enrolled patients with PVC's present prior to sedation with remifentanil IVPCA)
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Remifentanil: Remifentanil IV PCA
Arm/Group | Remifentanil
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 12
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Inhibition of Idiopathic Ventricular Tachycardia
Description: observation of the anesthetic effect on the inhibition of the ventricular tachycardia in patients undergoing radio-frequency ablation of idiopathic ventricular tachycardia. Patients were continuously monitored for presence of PVC's.
  Every 15 minutes patient's heart rhythm (EKG) was documented on the anesthetic record. Presence of PVC's of the same morphology was confirmed by the cardiologist performing the ablation.
Time Frame: duration of the procedure or until the presence of PVC's was no longer required for the cardiologist to complete the ablation, average 2 hours
Population: Study Data impacted by Storm Sandy in NYC and data lost for reporting
Arm/Group | Remifentanil IV PCA
Number analyzed (Participants) | 0

2. Primary Outcome: PVC Suppression With Remifentanil Sedation
Description: 1 observed suppression of PVC's (PVC's of the same morphology are no longer observed during any 15 minute recording interval) 0 no suppression
Time Frame: duration of the operative procedure, average 2 hours
Measure: Number; unit: participants with PVC suppression
Arm/Group | Remifentanil IV PCA
Number analyzed (Participants) | 16
participants with PVC suppression | 2
Statistical Analysis 1: Comparison: Remifentanil IV PCA; null hypothesis: Remifentanil IVPCA sedation in patients undergoing ablation of the idiopathic ventricular tachycardia does not cause suppression of PVC's; Test type: Superiority or Other; p = 0.05, Fisher Exact; Risk Difference (RD) = 0.65, 0.15% CI 2-sided [0.65 to 0.8], Standard Error of Mean 0.75

ADVERSE EVENTS:
Description: Serious and/or Other [non-serious] Adverse Events were not collected/assessed. Clinical sedation was provided in accordance with the standard of care adopted by the American Society of Anesthesiologists and approved by the medical center. Patients participating in the study were not at any additional risk.
Arm/Group | Remifentanil IV PCA
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No